CLINICAL TRIAL: NCT03542786
Title: Clinical Trial, Randomized and Controlled With Placebo to Evaluate the Addition to an Antiretroviral Treatment of a Probiotic, Only or in Conjunction of a Pre-biotical, in Adults Infected by Hiv-1 With a cd4 Record Less Than 500 Cells / mm3
Brief Title: Clinical Trial to Evaluate the Addition to an Antiretroviral Treatment of a Probiotic
Acronym: RECOVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Collaborators: Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I3.1 IRSICAIXA
Record Dates: First submitted 2018-05-08; First posted 2018-05-31 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: HIV; Premature Aging
Keywords: HIV-1
MeSH Terms: conditions — Aging, Premature | interventions — Probiotics; Prebiotics

STUDY DESIGN:
Intervention Model Description: 100 patients will be included in this trial. Patients will be randomized 2: 2: 1 to one of the following 3 branches according to the use of integrase inhibitors (INI), protease inhibitors (PI) or non-nucleoside analogue reverse transcriptase inhibitors ( ITINAN) and according to the CD4 count nadir is greater or less or equal to 200 cells / mm3: Branch A: add probiotic i3.1 to the antiretroviral therapy Branch B: add probiotic i3.1 and ProSeed prebiotic to the antiretroviral therapy Branch C: add placebo to ART The treatment periods will be of 6 months and follow-up will be carried out at month, at 3 months and at 6 after the start of the study treatment, and a last visit will be made at 3 months after discontinuing it (wash-out period).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- i3.1 (Experimental): This group will have their habitual antiretroviral therapy (integrase inhibitor (INI), protease inhibitor (IP), reverse transcriptase inhibitor (ITINAN)) combined with the research product (probiotic i3.1). The prebiotic will be taken once a day during 6 months.
  Interventions: Dietary Supplement: Probiotic
- i3.1 + ProSeed (Experimental): This group will have their habitual antiretroviral therapy combined with the probiotic (i3.1) and the prebiotic (ProSheed). The prebiotic and probiotic will be taken once a day during 6 months.
  Interventions: Dietary Supplement: Probiotic; Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): This group will only have their habitual antiretroviral therapy. The placebo will be taken once a day during 6 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The probiotic i3.1 is a commercialized product. It will be supplied by the promoter and manufactured in ALIFARM S.A.
  It contains:
  * Lactobacillus plantarum CECT7484
  * Lactobacillus plantarum CECT7485
  * Pediococcus acidilactici CECT7483
  Arms: i3.1; i3.1 + ProSeed
Dietary Supplement: Prebiotic — ProSeed prebiotic is a non-commercialized product. It will be supplied by the promoter and manufactured in ALIFARM S.A.
  It contains:
  * Partially Hydrolyzed Guar Gum (PHGG)
  * Inulin HPD
  * Oat Beta-Glucans
  * Pectin
  * Inulin Low Protein Diet (LPD)
  * Polydextrose
  * Maltrodextrins
  Arms: i3.1 + ProSeed
Dietary Supplement: Placebo — It is a non-commercialized product. It is composed of the same excipients as the probiotic and the prebiotic. It will be supplied by the promoter and manufactured in ALIFARM S.A.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate a therapy for the inflammaging (premature aging).

DETAILED DESCRIPTION:
It's been demonstrated that the HIV-1 virus is associated to the reduction of the microbiota. Some studies suggest that because of this bacterial reduction, the premature aging appears. So this study aims to demonstrate that our probiotic can balance the microbiota as a preventive solution for the inflammaging.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old.
* Documented HIV-1 infection.
* Be in treatment with these antiretrovirals (INI, IP, ITINAN) during 12 months.
* HIV-1 Viral titer <50 copies/mL during 6 months.
* CD4> 500 cells/mm3.

Exclusion Criteria:

* Treatment with antibiotics.
* Severe diseases actives.
* Defining diseases of AIDS in the previous year.
* Gut surgery except appendectomy or cholecystectomy.
* Pregnancy.
* Any diet deviation (vegans).
* Other probiotic treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
The appearance of adverse effects. | Change from Baseline Adverse Effects will be measured at 1 month and 3 months after the treatment beginning (V1 and V2 respectively).
  Percentage of patients with adverse events (AE) in the 3 study arms: i3.1, i3.1 + ProSeed and Placebo.

SECONDARY OUTCOMES:
Gut microbiota diversity and metabolomic profile | A measure will be made in V1, V2, V3 and V4 (1 month, 3 months, 6 months and 9 months after the treatment beginning, respectively).
  Biodiversity changes among the basal visit and 3 months after (in each arm), measured using the Shannon Index.
Translocational bacterial markers & Systemic inflammation markers | A measure will be made in V1 and V2 (1 month and 3 months after the treatment beginning, respectively).
  Markers changes among the basal visit and 3 months after, in each arm.The plasma levels of lipopolysaccharide, sCD14, Interleukin 6 and Iinterleukin 10 will be measured.
Cluster of Differentation 4 (CD4) count | A measure will be made in V2, V3 and V4 (3 months, 6 months and 9 months after the treatment beginning, respectively).
  Recount changes (cells/mm3) among the basal visit and 3 months after, in each arm.
CD4/CD8 ratio | A measure will be made in V2, V3 and V4 (3 months, 6 months and 9 months after the treatment beginning, respectively).
  Ratio changes among the basal visit and 3 months after, in each arm.
Satisfaction with the product | A measure will be made in V2, V3 and V4 (3 months, 6 months and 9 months after the treatment beginning, respectively).
  This parameter will be measured in order to evaluate the satisfaction of the patient with the research product. The satisfaction with the product wil be measured with the Likert Scale (with answers from satisfied to unsatisfied).
Questionaire to evaluate the life quality | A measure will be made in V2, V3 and V4 (3 months, 6 months and 9 months after the treatment beginning, respectively).
  This parameter will be measured with the Medical Outcomes Study-HIV questionaire (with answers from not affected to affected).
Questionaires to evaluate the anxiety and depression | A measure will be made in V2, V3 and V4 (3 months, 6 months and 9 months after the treatment beginning, respectively).
  This parameter will be measured with the Hospital Anxiety Depression Scale (HADS) questionaire (with answers from never to always).

CONTACTS AND LOCATIONS:
Overall Officials: Ariana Salavert, PhD, Study Director — AB-Biotics
Locations (1):
- Hospital Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blazquez-Bondia C, Parera M, Catala-Moll F, Casadella M, Elizalde-Torrent A, Aguilo M, Espadaler-Mazo J, Santos JR, Paredes R, Noguera-Julian M. Probiotic effects on immunity and microbiome in HIV-1 discordant patients. Front Immunol. 2022 Dec 8;13:1066036. doi: 10.3389/fimmu.2022.1066036. eCollection 2022. PMID 36569851